CLINICAL TRIAL: NCT04646304
Title: Motion Capture as a Tool for the Assessment of Laparoscopic Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 20200631-01H
Record Dates: First submitted 2020-11-03; First posted 2020-11-27 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Adult ALL
Keywords: surgical trainees; surgical staff
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Motion Capture

STUDY DESIGN:
Intervention Model Description: Phase 1 will recruit 4 groups of participants that vary in surgical experience (junior residents, senior residents, surgical fellows, and staff surgeons). Significant differences in objective measures of surgical performance will be identified. A target interval will be computed for each significant factor based on the staff surgeons' average performance.
  Phase 2 will recruit junior residents to complete the same sets of surgical tasks. Half of the participants will receive objective feedback comparing their performance in Set 1 to the staff surgeons' target interval while the other half will receive no feedback. Differences in performance between Sets 1 and 3 will be quantified and compared between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Objective Feedback (Motion Capture) (Other): Participants in the objective feedback group will receive a report that compares their performance in Set 1 to that of the staff surgeons' using the target interval as a reference. Participants receiving objective feedback will then complete Sets 2 and 3 knowing what factors to improve upon.
  Interventions: Other: Objective Feedback (Motion Capture)
- No Feedback (No Intervention): Participants receiving no feedback will complete all sets with no intervention.

INTERVENTIONS:
Other: Objective Feedback (Motion Capture) — Participants assigned to the objective feedback group will be given a report after completing Set 1 and Set 2. This report will outline their performance for each significant factor (identified in Phase 1) relative to a target interval, derived from the staff surgeon group average (± one standard deviation). Participants assigned to the objective feedback group will then be able to repeat the tasks knowing which variables to improve.
  Arms: Objective Feedback (Motion Capture)

SUMMARY:
The goal of this study is to 1) identify motion capture variables that can be used to differentiate surgical experience level and 2) evaluate if these variables can be used in a surgical education setting to improve resident performance.

DETAILED DESCRIPTION:
This will be a two-phase study that will take 2 years to complete.

Phase 1 will recruit staff surgeons, surgical fellows, and residents from the departments of Obstetrics and Gynecology, Urology, General Surgery, and Thoracics at The University of Ottawa and The Ottawa Hospital to complete a set of FLS tasks. Logistic regressions will be used to identify significant factors that differentiate surgical experience level (junior residents, senior residents, fellows, and staff). Classification of residents will depend on their current cohort in the CDB or traditional time-based system: A target interval will be computed for each significant factor based on the staff surgeons' average performance. This target interval will be used to assess resident performance in Phase 2.

Phase 2 will recruit Transition to Discipline residents from each department to complete 3 sets of FLS tasks. Participants will be randomized into an "objective feedback" group or a "no feedback" group. Participants randomized to the objective feedback group will receive a report that compares their performance in Set 1 to that of the staff surgeons' using the target interval as a reference. Participants receiving objective feedback will then complete Sets 2 and 3 knowing what factors to improve upon. Participants receiving no feedback will complete all sets with no intervention. Phase 2 data collection will start once Phase 1 is completed.

Trajectories of retro-reflective markers will be recorded using a 6-camera motion analysis system (40MXF-40 Vicon cameras, Oxford Metrics, Oxford, UK) sampling at 100 Hz with supporting Nexus software (v2, Oxford Metrics, Oxford, UK). Retro-reflective markers will be placed on various anatomical landmarks on the participant's body based on a cluster marker set. Laparoscopic surgical tools (grasper, scissors, or dissector) will have a marker triad fixed to the upper shaft while a laparoscopic trainer (FLS Trainer System, Limbs & Things, Savannah GA) will have markers placed at its corners. Using Vicon Nexus software, raw marker trajectories will be filtered and used to compute local coordinate systems of the upper body, joint centers, and subsequent joint angles while filtered marker trajectories on the laparoscopic tools will compute the tool tip's motion and orientation relative to the box trainer's workspace. Inertial measurement units (IMUs) will also be used to capture motion of the upper body and compare to motion capture outcomes (Secondary Objective). Wireless IMUs will be placed along the long axis of the forearm, upper arm, upper spine and lower spine.

Surface electromyography (EMG) signals of the biceps, triceps, anterior deltoid, upper trapezius, wrist extensors and flexors will also be recorded using a wireless EMG system (Trigno, Delsys Inc., Natick MA) and recorded using Nexus. Sensors will be placed over the muscle bellies following SENIAM guidelines [34] and signals will be sample data 100Hz with a 20-450Hz bandpass. All experimental EMG signals will be appropriately conditioned and normalized to maximum EMG value elicited during maximum voluntary isometric contraction (MVIC) exercises. Three repetitions of each MVIC exercise will be performed before the experimental task and will include elbow flexion and extension, arm abduction, arm flexion, and wrist flexion and extension. A minimum of 30 seconds rest will be given between each exercise to mitigate effects of fatigue.

Motion and EMG data will be exported to a custom MatLab (2019, Mathworks, Natick, MA) application to compute objective measures of laparoscopic performance: instrument tip pathlength, average (±1 stdev) excursion velocity, average (±1 stdev) excursion error, average (±1 stdev) upper body kinematics (shoulder, elbow, wrist, neck and trunk) in all three planes of motion, and integrated EMG.

Video of the surgical tasks will be recorded and synced to marker trajectory data using an external trigger. Videos will be de-identified, and the last repetition assessed by three staff surgeons. First, the raters will categorize each video as Transition to Discipline resident, Foundation of Discipline resident, Core Discipline resident, Transition to Practice resident, fellow, or staff surgeon based other their general perception of the performer's experience level. The raters will then score each video following the FLS scoring system (based on timing and penalty scores), and the OSATS evaluation grid.

ELIGIBILITY:
Inclusion Criteria:

* staff surgeons, surgical fellows and residents
* primary affiliation with the departments of Obstetrics and Gynecology, Urology, General Surgery, and Thoracics at the University of Ottawa and The Ottawa Hospital

Exclusion Criteria:

* current injury/condition that in the opinion or the participant and/or research team will affect performance

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Completion time | 1 year
  Time to complete each task measured in seconds
Instrument pathlength | 1 year
  Pathlength of surgical instrument tip measured in cm
Motion smoothness | 1 year
  Motion smoothness of surgical instrument tip measured by the number of changes in acceleration (m/s^2)
Instrument orientation | 1 year
  Orientation of surgical instrument tip measured in the three planes of motion (depth, pitch, roll, yaw), quantified in degrees relative to the surgical trainer box's local coordinate system.
Fundamentals of Laparoscopy Skill (FLS) score | 1 year
  - A numbered score is calculated following procedures outlined in the Fundamentals of Laparoscopy Skills (FLS) modules
Objective Structured Assessment of Technical Skills (OSATS) score | 1 year
  - A numbered score is computed from a global rating system based evaluation grid.
Participant classification | 1 year
  Blinded reviews will classify participants as junior residents, senior residents, fellows/staff based on their perception of participant skill level.

SECONDARY OUTCOMES:
Muscle Electromyography | 1 year
  * Muscles: erector spinae, biceps, triceps, anterior deltoid, upper trapezius, wrist extensors, wrist flexors
  * Amplitude quantified as %maximum measured during maximal effort trials
Muscle activation symmetry | 1 year
  * Muscles: erector spinae, biceps, triceps, anterior deltoid, upper trapezius, wrist extensors, wrist flexors
  * Symmetry indices will be quantified as non-dominant side/dominant side.
Upper body kinematics | 1 year
  - Body orientation will be measured in degrees for the shoulder, elbow, wrist, neck, trunk

CONTACTS AND LOCATIONS:
Overall Officials: Sukhbir Singh, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez A, Rodriguez O, Sanchez R, Benitez G, Pena R, Salamo O, Baez V. Laparoscopic surgery skills evaluation: analysis based on accelerometers. JSLS. 2014 Oct-Dec;18(4):e2014.00234. doi: 10.4293/JSLS.2014.00234. PMID 25489218
- [Background] Moorthy, Munz, Dosis, Bello, Darzi. Motion analysis in the training and assessment of minimally invasive surgery. Minim Invasive Ther Allied Technol. 2003 Jul;12(3):137-42. doi: 10.1080/13645700310011233. PMID 16754092
- [Background] Farcas MA, Trudeau MO, Nasr A, Gerstle JT, Carrillo B, Azzie G. Analysis of motion in laparoscopy: the deconstruction of an intra-corporeal suturing task. Surg Endosc. 2017 Aug;31(8):3130-3139. doi: 10.1007/s00464-016-5337-4. Epub 2016 Dec 7. PMID 27928669
- [Background] Gray RJ, Kahol K, Islam G, Smith M, Chapital A, Ferrara J. High-fidelity, low-cost, automated method to assess laparoscopic skills objectively. J Surg Educ. 2012 May-Jun;69(3):335-9. doi: 10.1016/j.jsurg.2011.10.014. PMID 22483134
- [Background] Ganni S, Botden SMBI, Chmarra M, Li M, Goossens RHM, Jakimowicz JJ. Validation of Motion Tracking Software for Evaluation of Surgical Performance in Laparoscopic Cholecystectomy. J Med Syst. 2020 Jan 24;44(3):56. doi: 10.1007/s10916-020-1525-9. PMID 31980955
- [Background] Gallagher AG, McClure N, McGuigan J, Ritchie K, Sheehy NP. An ergonomic analysis of the fulcrum effect in the acquisition of endoscopic skills. Endoscopy. 1998 Sep;30(7):617-20. doi: 10.1055/s-2007-1001366. PMID 9826140